CLINICAL TRIAL: NCT07405151
Title: A Phase 2 Open-Label, Umbrella Platform Design Study of Investigational Agent(s) in Participants With 2L/3L Unresectable Locally Advanced or Metastatic Esophageal Cancer: KEYMAKER-U06 Substudy 06F
Brief Title: A Clinical Trial of Ifinatamab Deruxtecan in People With Advanced Esophageal Cancer (MK-3475-06F)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-06F; 2025-524146-10 (Registry Identifier: EU CT); U1111-1329-6558 (Other: UTN); MK-3475-06F (Other: MSD)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Oesophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- I-DXd (Experimental): Participants will be administered I-DXd every 3 weeks until progressive disease or discontinuation criteria are met.
  Interventions: Biological: I-DXd; Drug: Rescue Medication

INTERVENTIONS:
Biological: I-DXd — IV Infusion
  Other Names: Ifinatamab Deruxtecan; DS-7300a; MK-2400
Drug: Rescue Medication — Includes 5-HT3 receptor antagonist, NK-1 receptor antagonist, and corticosteroid, administered per approved product label

SUMMARY:
The purpose of this trial is to assess if ifinatamab deruxtecan (I-DXd) can treat esophageal squamous cell carcinoma (ESCC). I-DXd is an antibody-drug conjugate (ADC). An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells.

The goal of this trial is to learn how many participants who receive I-DXd have the cancer respond, which means the cancer gets smaller or goes away.

DETAILED DESCRIPTION:
The master screening protocol is MK-3475-U06 (KEYMAKER-U06)

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of unresectable locally advanced or metastatic esophageal squamous cell carcinoma (ESCC)
* Has disease progression after 1 or 2 prior lines of systemic therapy for unresectable locally advanced or metastatic ESCC
* Has measurable disease
* If infected with human immunodeficiency virus (HIV), has well-controlled HIV on antiretroviral therapy
* Has adequate organ function

Exclusion Criteria:

* Has histologically or cytologically confirmed adenocarcinoma or adenosquamous carcinoma subtype
* Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention
* Has clinically significant corneal disease
* Has any of the following within 6 months before screening: cerebrovascular accident, transient ischemic attack, other arterial thromboembolic event
* If infected with HIV, has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has uncontrolled or significant cardiovascular disease
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has a history of (noninfectious) pneumonitis/interstitial lung disease irrespective of requiring steroids or has any current pneumonitis/interstitial lung disease or has suspected pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy other than those permitted.
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses, including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc), and potential pulmonary involvement caused by any autoimmune, connective tissue, or inflammatory disorders (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc), prior pneumonectomy, or requirement for supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-11 (Estimated); Primary Completion 2027-06-12 (Estimated); Study Completion 2028-06-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 15 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 18 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-Free Survival (PFS) | Up to approximately 18 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 27 months
  OS is defined as time from randomization to death due to any cause.
Number of Participants Who Experience an Adverse Events (AEs) | Up to approximately 18 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 18 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com